CLINICAL TRIAL: NCT04077762
Title: Radial Vs. State-Of-The-Art Femoral Access for Bleeding and Access SIte Complication Reduction in Cardiac Catheterization (REBIRTH)
Acronym: REBIRTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REBIRTH
Record Dates: First submitted 2019-08-26; First posted 2019-09-04 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Patient Satisfaction; Vascular Access Complication
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radial access (Active Comparator): Radial access for cardiac catheterization. Radial access will be performed using ultrasound guidance and a micropuncture needle or catheter-over-needle system, as per the local standard of care.
  Interventions: Procedure: Radial Access
- State-of-the-art femoral access (Active Comparator): Femoral access for cardiac catheterization. Femoral access will be obtained using state-of-the-art techniques (ultrasound and fluoroscopic guidance for arterial puncture, immediate femoral angiography after obtaining access and use of a vascular closure device whenever possible).
  Interventions: Procedure: State-of-the-art femoral access with 18 gauge needle; Procedure: State-of-the-art femoral access with 21 gauge needle

INTERVENTIONS:
Procedure: Radial Access — Radial Access
  Arms: Radial access
Procedure: State-of-the-art femoral access with 18 gauge needle — State-of-the-art femoral access with 18 gauge needle
  Arms: State-of-the-art femoral access
Procedure: State-of-the-art femoral access with 21 gauge needle — State-of-the-art femoral access with 21 gauge needle. For patients randomized to micropuncture (21G) the micropuncture wire must be advanced under fluoroscopy to avoid inadvertent wiring of side-branches.
  Arms: State-of-the-art femoral access

SUMMARY:
This is a phase IV, prospective, open label, randomized-controlled study that will compare radial access with state-of-the-art femoral access in patients without ST-segment elevation acute myocardial infarction undergoing cardiac catheterization. Subjects will be randomized 1:1 into 2 treatment groups: radial access and state-of-the-art femoral access. Randomization will be performed in blocks of 50 per site. Similarly, a second sub-randomization will be performed in the femoral access group into use of 18 vs 21 gauge needles, also in a 1:1 fashion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Undergoing diagnostic angiography for ischemic symptoms with possible PCI, or undergoing planned urgent or elective PCI
* Has provided informed consent and agrees to participate
* Patients must be equally eligible to undergo cardiac catheterization via radial or femoral access

Exclusion Criteria:

* Primary PCI for STEMI
* Planned right heart catheterization
* Valvular heart disease requiring valve surgery within 30 days after the index procedure
* Hemodialysis access (arteriovenous fistula or graft) in the arm to be used for PCI in case of assignment to radial approach (the opposite arm may be used for radial access if a dialysis graft is present in one)
* Peripheral arterial disease prohibiting vascular access
* Presence of bilateral internal mammary artery coronary bypass grafts
* International normalized ratio ≥1.5 while treated with oral vitamin K antagonists (i.e. warfarin) Receipt of oral factor Xa or IIa inhibitors ≤24 h before procedure
* Planned staged PCI within 30 days after index procedure.
* Any planned surgeries within 30 days after index procedure
* Planned dual arterial access (for example for chronic total occlusion PCI)
* Coexisting conditions that limit life expectancy to less than 30 days
* Positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3266 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2027-08-19 (Estimated); Study Completion 2028-08-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite of vascular access complications and bleeding (BARC 2, 3, or 5) | Evaluations will occur up to 30 days

SECONDARY OUTCOMES:
Total number of BARC type 2, 3, or 5 bleeding events | Evaluations will occur up to 30 days
Number of Vascular access complications defined as the composite of arteriovenous fistula, arterial pseudoaneurysm, or arterial occlusion requiring intervention; | Evaluations will occur up to 30 days
Number of participants with Radial artery occlusion | Evaluations will occur up to 30 days
Number of participants with Access site crossover | Measured during procedure
  The inability to complete the procedure from the assigned arterial access site, requiring conversion from radial to femoral access or vice versa for procedure completion
Number of other vascular access related complications | Evaluations will occur up to 30 days
Total procedure time | Measured during procedure
  The time from administration of local anesthesia to the time of removal of all interventional equipment
Time to ambulation | Measured up to 24 hours after procedure completion
Number of all cause death and cardiac death | Evaluations will occur up to 30 days
Number of participants with Myocardial Infarction | Evaluations will occur up to 30 days
  The 4th Universal Definition of myocardial infarction
Number of participants with Stroke | Evaluations will occur up to 30 days
Number of participants with unplanned coronary revascularization | Evaluations will occur up to 30 days
Measure of Radiation Dose | Measured during procedure
  Both air kerma and dose air product
Fluoroscopy Time | Measured during procedure
Contrast volume | Measured during procedure
Number of participants with Procedural Success | Evaluations will occur up to 30 days
  Using the National Cardiovascular Disease Registry (NCDR) definition
Duration of hospital stay and frequency of same day discharge | Evaluations will occur up to 30 days
Patient Preference Survey: Radial Vs Femoral Access | Evaluations will occur up to 30 days
  Participants will be asked which access site they would have preferred to have their procedure

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil Brilakis, MD, PhD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (6):
- United States (6):
  - San Francisco VA Medical Center, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Joseph Maxwell Cleland Atlanta VA Medical Center, Decatur, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140